CLINICAL TRIAL: NCT02138279
Title: Comparative Study of the Topcon Tonometers - CT-800, CT-1, CT-1P and TRK-2P to Demonstrate Conformance to ANSI Z80.10-2009 Ophthalmic Instruments -Tonometers, to the FDA Guidance for Industry and FDA Staff, Tonometer-Premarket Notification [510(k)] Submissions, and to the Applicable Supplemental Information Sheet and Comparison of Pachymetry Values for CT-1P and TRK-2P With the Konan CellChek Plus (Predicate)
Brief Title: Comparative Study of Non-contact Tonometers for Intraocular Pressure and Corneal Cell Thickness Measurements
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: TOPCON-TON-US-0001
Record Dates: First submitted 2014-04-23; First posted 2014-05-14 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Intraocular Pressure; Corneal Pachymetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Male and female adults 18+ years of age

SUMMARY:
The primary objective of this clinical study is to collect clinical data to support FDA 510(k) submissions for the Topcon CT-800, CT-1, CT-1P and TRK-2P non-contact tonometers. The secondary objective is to evaluate any adverse events found during the clinical study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age of either sex and any race or ethnicity;
* Willing and able to provide written informed consent prior to any study procedures being performed;
* Willing and able to follow all instructions and attend all study visits;
* Best Spectacle Corrected Visual Acuity (BSCVA) of 0.3 logMAR (20/40 Snellen equivalent) or better in both eyes as measured using an ETDRS chart.

Exclusion Criteria:

* Only one functional eye;
* Poor or eccentric fixation;
* Corneal scarring or have had corneal surgery, including corneal laser surgery;
* Microphthalmos;
* Buphthalmos;
* Contact lens wearer, meaning having worn soft contact lenses within the past 3 months and/or rigid permeable gas lenses within the past 6 months;
* Dry eyes, meaning having been diagnoses by a physician with dry eyes and currently using a prescribed medication;
* Lid squeezer - blepharospasm;
* Nystagmus;
* Keratoconus;
* Any other corneal or conjunctival pathology or infection;
* Condition or a situation, which in the Investigator's opinion, may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ophthalmology practice
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Agreement of intraocular pressure measurements from predicate vs. investigational device | Single timepoint - 1 day
Agreement of central corneal thickness measurements from predicate vs. investigational device | Single time point - 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States